CLINICAL TRIAL: NCT03510910
Title: Multimodal Analgesia With Acetaminophen vs. Narcotics Alone After Hip Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00167
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Hip Arthroscopy
MeSH Terms: interventions — Acetaminophen; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acetaminophen along with a reduced quantity of Percocet (Experimental)
  Interventions: Drug: Acetaminophen; Drug: Percocet
- Percocet only (Experimental)
  Interventions: Drug: Percocet

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen 600 mg to be taken every 8 hours (TID)
  Arms: Acetaminophen along with a reduced quantity of Percocet
Drug: Percocet — Oxycodone/acetaminophen (Percocet) 5 mg/325 mg as needed for breakthrough pain for patients in Percocet+ Acetaminophen group.
  Percocet Group will receive standard of care Percocet 5 mg/325 mg every 6 hours PRN

SUMMARY:
The purpose of this proposed study is to evaluate the efficacy of a multimodal approach to analgesia for patient's pain after hip arthroscopy and to also assess if this new approach will result in a reduction in post-operative narcotic use.

This study is a single-center, randomized prospective study comparing post-operative pain scores and narcotic consumption between individuals receiving acetaminophen along with a reduced quantity of Percocet (to be used as needed for breakthrough pain) and individuals receiving Percocet only. Both pain management options are considered to be standard of care. Both cohorts will receive aspirin for DVT prophylaxis and celecoxib for heterotopic ossification prophylaxis.

The primary objective of the study are to compare patients' narcotic consumption and reported pain following arthroscopic hip surgery, and determine if acetaminophen can provide adequate pain relief compared to a narcotic medication.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II
* Patients indicated and scheduled for arthroscopic hip surgery

Exclusion Criteria:

* Contraindication to acetaminophen or oxycodone/acetaminophen (e.g. hypersensitivity, history of GI or bleeding disorder)
* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age or older than 65
* Any patient considered a vulnerable subject
* Patients on pain medication prior to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Youm, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen Along With a Reduced Quantity of Percocet: Acetaminophen: acetaminophen 600 mg to be taken every 8 hours (TID)
  Percocet: Oxycodone/acetaminophen (Percocet) 5 mg/325 mg as needed for breakthrough pain for patients in Percocet+ Acetaminophen group.
  Percocet Group will receive standard of care Percocet 5 mg/325 mg every 6 hours PRN
Period: Overall Study
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
Started | 42 | 43
Completed | 40 | 40
Not Completed | 2 | 3
Not completed — Incomplete Survey | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Standard Deviation); unit: years] | 39.43 (13.1) | 40.2 (16.5) | 39.82 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 16 | 18 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Satisfaction was reported on a Likert-type scale of 1-10 (the higher the score, the higher the satisfaction)
Time Frame: 7 days post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
Number analyzed (Participants) | 40 | 40
score on a scale | 8.48 (1.52) | 8.83 (1.55)

2. Primary Outcome: Morphine-equivalent Consumption
Description: Amount of oxycodone/acetaminophen (Percocet) in 5mg/325mg doses will be recorded in number of pills
Time Frame: 7 days post-surgery
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
Number analyzed (Participants) | 40 | 40
pills | 6.33 (7.1) | 5.69 (5.8)

3. Primary Outcome: Score on Visual Analog Scale (VAS) of Pain
Description: Pain severity scores at rest will be assessed by use of VAS. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The higher the score, the worse the pain.
Time Frame: 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
Number analyzed (Participants) | 40 | 40
score on a scale | 5.30 (2.02) | 4.98 (2.24)

4. Primary Outcome: Score on Visual Analog Scale (VAS) of Pain
Description: as for outcome 3
Time Frame: 4 days post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
Number analyzed (Participants) | 40 | 40
score on a scale | 3.55 (1.68) | 3.20 (1.98)

5. Primary Outcome: Score on Visual Analog Scale (VAS) of Pain
Description: as for outcome 3
Time Frame: 7 days post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
Number analyzed (Participants) | 40 | 40
score on a scale | 3.20 (1.79) | 2.83 (2.11)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Acetaminophen Along With a Reduced Quantity of Percocet | Percocet Only
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03510910/Prot_SAP_000.pdf